CLINICAL TRIAL: NCT04622696
Title: A Post-market Clinical Follow-up Study to Evaluate the Safety and Performance of the HydroMARK® Breast Biopsy Site Marker
Brief Title: HydroMARK Post-market Clinical Follow-up Study
Status: Completed | Type: Observational
Sponsor: Devicor Medical Products, Inc. (Industry)
Responsible Party: Sponsor
Organization: Leica Biosystems (Industry)
Other Study IDs: LBS-CA-PTL-033
Record Dates: First submitted 2020-10-26; First posted 2020-11-10 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer
Keywords: Radiology; Breast Biopsy; Ultrasound visibility
MeSH Terms: conditions — Breast Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Prospective - Performance Cohort: Subjects will undergo an ultrasound-guided breast biopsy procedure with placement of HydroMARK Breast Biopsy Site Marker per site standard of care and will return to the office at 6-12 weeks post-implant for ultrasound imaging to evaluate device visibility.
  Interventions: Diagnostic Test: Ultrasound imaging
- Retrospective - Safety Cohort: Device-related adverse events will be collected via retrospective medical chart review for a minimum of 90 days post-HydroMARK Breast Biopsy Site Marker implant (unless the subject was exited according to the medical records due to the implant being removed/explanted or subject death).

INTERVENTIONS:
Diagnostic Test: Ultrasound imaging — Subjects in the performance cohort will undergo ultrasound imaging to assess the visibility of the HydroMARK Breast Biopsy Marker at 6-12 weeks post-implant. There is no intervention in the safety cohort (retrospective chart review).
  Groups: Prospective - Performance Cohort

SUMMARY:
The purpose of this study is to assess the safety and performance of the HydroMARK Breast Biopsy Site Marker manufactured in the Devicor Medical Products, Inc. Tijuana facility.

ELIGIBILITY:
Inclusion Criteria:

Safety Cohort

* Subject was implanted during a breast biopsy procedure with a HydroMARK Breast Biopsy Site Marker manufactured at the Devicor Tijuana facility per the instructions for use
* Subject has been followed at least 90 days according to the hospital's standard of care (SOC)
* Subject was ≥ 18 years of age at the time of the breast biopsy procedure
* Subject has accessible medical records documenting the breast biopsy procedure including, at minimum: age, sex, primary diagnostic indication and documentation of device-related adverse events which occurred, if any

Performance Cohort

* Subject was implanted during a breast biopsy procedure with a HydroMARK Breast Biopsy Site Marker manufactured at the Devicor Tijuana facility per the instructions for use
* Patient is ≥18 years of age
* Patient has provided informed consent to participate in study, including follow-up visit for ultrasound imaging at 6-12 weeks post-biopsy

Exclusion Criteria:

Safety Cohort

• Biopsy area was infected at the time of implant

Performance Cohort

* Contraindication to HydroMARK Breast Biopsy Site Marker implantation
* Biopsy area is infected at the time of implant
* Patient has a breast biopsy marker (in the same breast) implanted from a previous procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Safety cohort: retrospective chart review of ~491 subjects who underwent a breast biopsy procedure with implant of a HydroMARK Breast Biopsy Site Marker manufactured at the Devicor Tijuana facility.
  Performance cohort: ~341 subjects with a suspected breast cancer that will undergo as part of standard of care an ultrasound-guided breast biopsy procedure, including placement of HydroMARK Breast Biopsy Site Marker manufactured at the Devicor Tijuana facility, with an aim of achieving a minimum 239 evaluable subjects returning to the office at 6-12 weeks for ultrasound imaging to evaluate device visibility.
Sampling Method: Non-Probability Sample
Enrollment: 730 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
Safety Cohort | 90 days post-implant
  The safety cohort will consist of approximately 491 evaluable subject medical records reviewed retrospectively from patients followed for a minimum of 90 days post-implant unless the subject was exited according to the medical records due to the implant being removed/explanted or subject death. Device-related adverse events and device deficiencies will be collected.
Performance Cohort | 6 - 12 weeks post-implant
  The performance cohort will prospectively enroll approximately 341 subjects with a suspected breast cancer that will undergo as part of standard of care an ultrasound-guided breast biopsy procedure, including placement of HydroMARK, with an aim of achieving a minimum 239 evaluable subjects (assuming 30% attrition rate due to surgical excision prior to follow-up, lost to follow-up, death) returning to the office at 6-12 weeks for ultrasound imaging to evaluate HydroMARK visibility.
  The visibility rate will be dichotomized into two categories from rankings using a 1-5 Likert-type scale - 1 "no/inadequate visibility" and 2 "slightly visible", 3 "moderately visible", 4 "very visible" and 5 "extremely visible" will be coalesced into a single category of "being visible".

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - ProMedica Toledo Hopsital, Toledo, Ohio
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No